CLINICAL TRIAL: NCT05082857
Title: Pediatric Parenting Connections Young Moms Program
Brief Title: (YMP) Young Moms Program
Acronym: YMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00076601; UL1TR001420 (NIH)
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Chronic Toxic Stress; Developmental/ Behavioral Regression in Young Children
Keywords: young moms; child health; teen births; child maltreatment; food insecurity

STUDY DESIGN:
Intervention Model Description: The study team will employ a blind randomized design to assign individuals to either the "traditional" Parents as Teachers (PAT) or the "hybrid" PAT model.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "traditional" Parents as Teachers (PAT) (Active Comparator): A twice-a-month home visits from trained family educators. Home visits will continue for the remainder of the study period as will the other components of the Parents as Teachers model: regular Group Connections for peer interactions and support, age-appropriate health and developmental screenings, and referrals that reflect mother and infant needs to community agencies that include the Child Development Services Agency (which provides screening for Individuals with Disabilities in Education Act (IDEA) Part C services), family services, intensive mental health services, among others. The study team will collect baseline data during the first home visit and complete monthly questionnaires during each month the mother is enrolled. An outcome assessment and participation in a focus group will be administered the last month of the study.
  Interventions: Behavioral: "traditional" Parents as Teachers (PAT)
- "hybrid" PAT model (Experimental): A six-week virtual evidence-based parenting class entitled What You Do Matters, which will be delivered in partnership with the Pediatric Advocacy Program at WFBMC which combines short parent-educator discussions followed by interactive activities and peer to peer networking. Young moms will participate in Group Connections for peer interactions and support. After completing the six-week course, teens will begin receiving once a month home visits, ongoing Group Connections, age-appropriate health and developmental screenings, and referrals that reflect mother and infant needs to other community agencies and resources, as listed above. The study team will collect baseline data prior to the beginning of the virtual What You Do Matters program and will complete monthly questionnaires during each month the mother is enrolled. An outcome assessment and participation in a focus group will be administered the last month of the study.
  Interventions: Behavioral: "hybrid" PAT model

INTERVENTIONS:
Behavioral: "traditional" Parents as Teachers (PAT) — A twice-a-month home visits from trained family educators. Home visits will continue for the remainder of the study period as will the other components of the Parents as Teachers model: regular Group Connections for peer interactions and support, age-appropriate health and developmental screenings, and referrals that reflect mother and infant needs to community agencies that include the Child Development Services Agency (which provides screening for Individuals with Disabilities in Education Act (IDEA) Part C services), family services, intensive mental health services, among others.
  Arms: "traditional" Parents as Teachers (PAT)
Behavioral: "hybrid" PAT model — A six-week virtual evidence-based parenting class entitled What You Do Matters, which will be delivered in partnership with the Pediatric Advocacy Program at WFBMC which combines short parent-educator discussions followed by interactive activities and peer to peer networking.
  Arms: "hybrid" PAT model

SUMMARY:
Young Moms Program (YMP) is designed to address systemic barriers to the health and stability of young moms and their children such as the lack of coordination of service delivery or logistical barriers within the health system. The YMP also streamlines the referral pipeline, connecting moms to evidence-based resources, and ensuring children complete all recommended assessments prior to kindergarten.

DETAILED DESCRIPTION:
This application is a community-engaged research collaboration between the non-profit Imprints Cares, the Wake Forest Baptist Medical Center (WFBMC) Birth Center, and Wake Forest School of Medicine (WFSOM). This project addresses the myriad risks associated with young moms ≤ 21 years old. Because YMP is a tiered program model, services meet parents where they are through a "warm hand-off" approach that uses one-on-one consultation and assessment-based interventions.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be an immediately post-partum mother
* Subject will reside with her newborn
* Subject must be referred from either the Birth Center at Wake Forest Baptist Health or from one of the Wake Forest Baptist Health Patient Priorities Care (PPC) partner practices
* Participants must speak English or Spanish

Exclusion Criteria:

* Newborn of participating mothers must be >= 35 weeks of gestation and not have an extended neonatal intensive care unit (NICU) stay

Ages: 14 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — outcome measures are only applicable to female participants
Enrollment: 15 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Miller-Fitzwater, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Science, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 screen failures prior to randomization
Period: Overall Study
Arm/Group | "Traditional" Parents as Teachers (PAT) | "Hybrid" PAT Model
Started | 6 | 9
Completed | 3 | 5
Not Completed | 3 | 4
Not completed — participants relocated and could not continue | 2 | 1
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: 6 participants who screen failed are not included in baseline characteristics
Groups:
- Total: Total of all reporting groups
Arm/Group | "Traditional" Parents as Teachers (PAT) | "Hybrid" PAT Model | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.33 (1.8) | 20.22 (1) | 19.9 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Protective Factors Survey Score
Description: The Protective Factors Survey (PFS) is a 20-item measure - The PFS is a validated parent survey designed that assesses protective factors in five areas: family functioning/resiliency, social emotional support, concrete support, nurturing and attachment, and knowledge of parenting/child development - Each subscale is rated 1-7; higher is better - range is 35-175
Time Frame: Week 1
Population: One Traditional model patient did not complete the PFS at 1 week (but completed all of the other items) and there was a drop out of a hybrid patient by the 6 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 9 | 5
score on a scale | 104.7 (12.7) | 98 (4.7)

2. Primary Outcome: Protective Factors Survey Score
Description: as for outcome 1
Time Frame: Week 6
Population: One Traditional model patient did not complete the PFS at 1 week (but completed all of the other items) and there was a drop out of a hybrid patient by the 6 week. The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 8 | 6
score on a scale | 104.1 (10) | 101.8 (7.9)

3. Primary Outcome: Protective Factors Survey Score
Description: as for outcome 1
Time Frame: Month 6
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 5 | 3
score on a scale | 108 (6.8) | 104.7 (14)

4. Primary Outcome: Number of Children Screen Positive for Delays Using the Ages and Stages Questionnaire (ASQ 3) Score
Description: The Ages and Stages Questionnaire (ASQ 3) is a validated developmental screening designed for use by and with parents. The ASQ 3 screens for developmental milestones in communication, gross motor, fine motor, problem solving, and personal-social skills - Range is 0-60 for all age levels, higher is better
Time Frame: Month 2
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Number; unit: number of participants
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 8 | 6
number of participants | 1 | 0

5. Primary Outcome: Number of Children Screen Positive for Delays Using the Ages and Stages Questionnaire (ASQ 3)
Description: as for outcome 4
Time Frame: Month 4
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Number; unit: number of participants
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 5 | 4
number of participants | 0 | 1

6. Primary Outcome: Number of Children Screen Positive for Delays Using the Ages and Stages Questionnaire (ASQ 3)
Description: as for outcome 4
Time Frame: Month 6
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Number; unit: number of participants
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 5 | 3
number of participants | 0 | 0

7. Primary Outcome: Number of Children Screen Positive for Delays Using the Ages and Stages Questionnaire: Social-Emotional (ASQ:SE 2) Score
Description: The Ages and Stages Questionnaire: Social-Emotional (ASQ:SE 2) is a validated screening of social and emotional behaviors - Range 0-240, Monitor with scores 25-34, score positive and refer with scores >=35
Time Frame: Month 2
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Number; unit: number of participants
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 8 | 6
number of participants | 0 | 0

8. Primary Outcome: Number of Children Screen Positive for Delays Using the Ages and Stages Questionnaire: Social-Emotional (ASQ:SE 2) Score
Description: The Ages and Stages Questionnaire: Social-Emotional (ASQ:SE 2) is a validated screening of social and emotional behaviors - Range 0-345, Monitor with scores 35-44 , score positive and refer with scores >=45
Time Frame: Month 6
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Number; unit: number of participants
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 5 | 3
number of participants | 0 | 0

9. Primary Outcome: The Patient Health Questionnaire (PHQ 9) Score
Description: The Patient Health Questionnaire (PHQ 9) is a self-administered questionnaire that is validated for use in assessing the severity of depression.
  Depression Severity: 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe. Validity has been assessed against an independent structured mental health professional (MHP) interview. PHQ-9 score ≥10 had a sensitivity of 88% and a specificity of 88% for major depression.
Time Frame: Baseline
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 9 | 6
score on a scale | 2.2 (2.7) | 3.8 (4.2)

10. Primary Outcome: The Patient Health Questionnaire (PHQ 9) Score
Description: as for outcome 9
Time Frame: Month 6
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 5 | 3
score on a scale | 4.6 (6.0) | 3.3 (3.5)

11. Primary Outcome: The StimQ2-I Infant Cognitive Home Environment Questionnaire Score No Availability of Learning (ALM)
Description: The StimQ2-I is a validated, interview-based assessment of home environments for use with infants ages five to 12 months. The StimQ2-I focuses on cognitive stimulation by the primary caregiver and contains several scales: Reading-Verbal, Parental Involvement in Developmental Advance, and Parental Verbal Responsivity - subscale range Read = 15, Parental Involvement in Developmental Advance (PIDA) = 5, Performance Validity Test (PVT) = 16 -Total STIMQ-I score range for the no ALM portion is 0-36; higher score is better.
Time Frame: Month 6
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 5 | 3
score on a scale | 29.4 (4) | 20.3 (11.1)

12. Primary Outcome: Full STIMQ2-I Including Availability of Learning Materials (ALM)
Description: The StimQ2-I is a validated, interview-based assessment of home environments for use with infants ages five to 12 months. The StimQ2-I focuses on cognitive stimulation by the primary caregiver and contains several scales: Availability of Learning Materials, Reading-Verbal, Parental Involvement in Developmental Advance, and Parental Verbal Responsivity - subscale range Read = 15, Parental Involvement in Developmental Advance (PIDA) = 5, Performance Validity Test (PVT) = 16, Availability of Learning Materials (ALM) = 6 Total score range for the STIMQ2-I including ALM is 0-42--a higher score is better.
Time Frame: Month 6
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 5 | 3
score on a scale | 40.4 (11.10) | 28 (11.14)

13. Secondary Outcome: Percent of Mothers Currently Using Contraception
Description: Percent of participants regularly using effective contraception
Time Frame: Month 6
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Number; unit: percentage of mothers
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 5 | 3
percentage of mothers | 60 | 67

14. Secondary Outcome: Percent of Mothers Breastfeeding
Description: Percent of mothers breastfeeding
Time Frame: Week 6, Month 3 and Month 6
Population: Data not collected at week 6 for any participant. The data was not collected for each outcome for participants missing from the numbers analyzed in each arm.
Measure: Number; unit: percentage of mothers
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 9 | 6
percentage of mothers
  Week 6: number analyzed (Participants) | 0 | 0
  Month 3: number analyzed (Participants) | 6 | 4
  Month 3 | 80 | 50
  Month 6: number analyzed (Participants) | 5 | 3
  Month 6 | 60 | 0

15. Secondary Outcome: Number of Completed Well Child Visits
Description: The team will track completion of well-child visits
Time Frame: Week 1, Months 2, 4, and 6
Population: Data not collected for this outcome
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Number of Completed Immunizations
Description: The team will track completion of immunizations
Time Frame: Months 2, 4, and 6
Population: Data not collected for this outcome.
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Number of Emergency Department (ED) Visits Per Subject
Description: The team will use WFBMC Epic data to track use of preventive rather than emergent health care
Time Frame: Month 6
Population: Data not collected for this outcome
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Percent of Mothers That Continue Current Educational Pathway
Description: The study team will track whether or not participants continue their education during the study period
Time Frame: Month 6
Population: The data was not collected for this outcome for participants missing from the numbers analyzed in each arm.
Measure: Number; unit: percentage of mothers
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 5 | 3
percentage of mothers | 20 | 33

19. Secondary Outcome: Number of Referrals Placed Per Subject
Description: Program services include developmental screenings, which in turn can lead to diagnostic assessments and, when eligible, enrollment in services. The team will track those infants are receiving the recommended screenings in a timely manner. Then, in cases where there are concerns, the team will follow-up with the young mom to determine whether or not the parent completed a formal assessment and, if eligible, enrolled in services.
Time Frame: Month 6
Population: Data not collected for this outcome
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Percent of Referrals Completed
Description: as for outcome 19
Time Frame: Month 6
Population: Data not collected for this outcome measure
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Percent of Completed Referrals That Result in Services
Description: as for outcome 19
Time Frame: Month 6
Population: Data not collected for this outcome measure
Arm/Group | "Hybrid" PAT Model | "Traditional" Parents as Teachers (PAT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline through month 6
Arm/Group | "Traditional" Parents as Teachers (PAT) | "Hybrid" PAT Model
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 0/6 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT05082857/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT05082857/ICF_000.pdf